CLINICAL TRIAL: NCT04802109
Title: The Impact of Rescuer Fatigue and Quality During Cardiopulmonary Resuscitation by Using Personal Protective Equipment. A Randomized Controlled Crossover Trial.
Brief Title: The Rescuer Fatigue During Cardiopulmonary Resuscitation in Manikin by Using Personal Protective Equipment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: An-Nan Hospital, China Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: TMANH109-REC017
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Cardiac Arrest
Keywords: personal protective equipment; rescuer fatigue; N-95; Powered Air-Purifying Respiratory
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective randomized crossover trial . Each participant is required to perform a five-minute CPR in kneeling position using three different types of personal protective equipment. After each round of CPR for 5 minutes, the participants can rest for two hours before the next round of CPR with different type of personal protective equipment
Who Masked: Outcomes Assessor
Masking Description: It is impossible to masking the participant, care provider during the CPR study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPR with level D PPE (Placebo Comparator): The participant doing CPR for 5 minutes with wearing level D personal protective equipment with surgical face mask
  Interventions: Device: wearing level D personal protective equipment; Device: wearing Level C personal protective equipment with N-95; Device: wearing Level C personal protective equipment with Powered Air-Purifying Respiratory
- CPR with level C PPE (Experimental): The participant doing CPR for 5 minutes with Level C personal protective equipment with N-95 face mask
  Interventions: Device: wearing level D personal protective equipment; Device: wearing Level C personal protective equipment with N-95; Device: wearing Level C personal protective equipment with Powered Air-Purifying Respiratory
- CPR with Level C PPE + PAPR (Experimental): The participant doing CPR for 5 minutes with Level C personal protective equipment with Powered Air-Purifying Respiratory.
  Interventions: Device: wearing level D personal protective equipment; Device: wearing Level C personal protective equipment with N-95; Device: wearing Level C personal protective equipment with Powered Air-Purifying Respiratory

INTERVENTIONS:
Device: wearing level D personal protective equipment — rubber gloves + surgical face mask + general isolation clothing
Device: wearing Level C personal protective equipment with N-95 — C-level protective clothing+ N95 mask + disposable protective clothing ("Ten Quin" Medial Apparel) + foot cover + rubber gloves + mask + general isolation clothing
Device: wearing Level C personal protective equipment with Powered Air-Purifying Respiratory — C-level protective clothing+ N95 mask + disposable protective clothing ("Ten Quin" Medial Apparel) + foot cover + rubber gloves + mask + general isolation clothing+Powered Air-Purifying Respiratory

SUMMARY:
Background:

High-quality cardiopulmonary resuscitation is the key to recovering patients with sudden cardiac death. However, when the environment is exposure to biologic hazard, the medical personnel need to use different personal protective equipment while doing CPR, and this difficulty is greatly increased. The research on this part is quite limited, and the results need to be further analyzed.

Purpose:

Compare the effects of CPR wearing different levels of personal protective equipment on CPR quality and rescue fatigue.

Material & Methods:

This study is designed as a prospective randomized crossover trial with an expected total of 40 volunteer participants, performed during 2021 April 1 to 2021 June 30. Each participant is required to perform a five-minute CPR in kneeling position using three different types of personal protective equipment. These three modes are Level D protective equipment with surgical mask, Level C protective equipment with N-95 mask, and Level-C protective equipment with Powered Air Purifying Respirator. Participants are physicians or nurses at the hospital. The participation are randomly assigned to the order of the three modes, and each mode can be rested for 120 minutes. Laerdal Skillreporter is used for CPR and quality measurement. The main results were effective chest compression ratio, correct chest depth ratio, correct chest recoil ratio and chest compression number per minute. The secondary results were personal blood pressure before and after the CPR, heartbeat, pulse oximeter, number of breaths, and subjective fatigue index (VAS 1 ~ 100 points), Questionnaire for the opinion of wearing personal protective equipment and using the porta count test to test the N-95 face mask for its quantitative fitness factor before and during CPR, and infrared detector for qualitative fitness test.

DETAILED DESCRIPTION:
Background:

High-quality cardiopulmonary resuscitation is the key to recovering patients with sudden cardiac death. However, when the environment is exposure to biologic hazard, the medical personnel need to use different personal protective equipment while doing CPR, and this difficulty is greatly increased. The research on this part is quite limited, and the results need to be further analyzed.

Purpose:

Compare the effects of CPR wearing different levels of personal protective equipment on CPR quality and rescue fatigue.

Material & Methods:

This study is designed as a prospective randomized crossover trial with an expected total of 40 volunteer participants, performed during 2021 April 1 to 2021 June 30. Each participant is required to perform a five-minute CPR in kneeling position using three different types of personal protective equipment. These three modes are Level D protective equipment with surgical mask, Level C protective equipment with N-95 mask, and Level-C protective equipment with Powered Air Purifying Respirator. Participants are physicians or nurses at the hospital. The participation are randomly assigned to the order of the three modes, and each mode can be rested for 120 minutes. Laerdal Skillreporter is used for CPR and quality measurement. The main results were effective chest compression ratio, correct chest depth ratio, correct chest recoil ratio and chest compression number per minute. The secondary results were personal blood pressure before and after the CPR, heartbeat, pulse oximeter, number of breaths, and subjective fatigue index (VAS 1 ~ 100 points), Questionnaire for the opinion of wearing personal protective equipment and using the porta count test to test the N-95 face mask for its quantitative fitness factor before and during CPR, and infrared detector for qualitative fitness test.

Inclusion criteria:

physicians and nurses from An Nan Hospital, with more than one year of work experience, possessing ACLS or BLS certificate, regardless of gender, height and weight.

Exclusion criteria:

back pain in the past, spine surgery, sciatica, coronary heart disease, and lung diseases such as asthma or chronic obstructive pulmonary disease. Pregnant women need to be excluded.

Statistic Method On the basis of our previous study (Foo NP,et al.Rescuer fatigue and cardiopulmonary resuscitation positions: A randomized controlled crossover trial. Resuscitation. 2010;81(5):579-584). we estimated that with a level of 0.05, a power of 80%, and an effect size of 0.6, a sample size of 18 participants would be sufficient for evaluating the primary outcome. We applied the Shapiro-Wilk test to evaluate the normality of the distribution of data. Then, we applied ANOVA for repeat measures and the Bonferroni procedure to evaluate the differences among and between different positions if the data fit the Gaussian distribution, and the Friedman test and Wilcoxon signed rank test if the data did not fit the Gaussian distribution. All the statistical tests were performed at the two-tailed level of significance at 0.05, and all statistical analyses were performed using SPSS for Windows, Version 17.0 (SPSS Inc., Chicago, U.S.A.).

ELIGIBILITY:
Inclusion Criteria:

* Physicians and nurses at An Nan Hospital, with more than one year of work experience, with Advanced cardiac life support or basic life support certificate

Exclusion Criteria:

* back pain in the past, spine surgery, sciatica, coronary heart disease, and lung diseases such as asthma or chronic obstructive pulmonary disease. Pregnant women are also excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
effective chest compression ratio | 5 minutes
  each chest compression that deep greater than 5 cm, around 100~120 times per minutes and recoil during each chest compression

SECONDARY OUTCOMES:
quantitative fitness factor of face mask | 5 minutes
  using porta count to detect the quantitative fitness factor of face mask. data from 0~200, if >=100 remain qualified outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ning-Ping Foo, PhD, Study Director — Director of Department of Emergency Medicine
Locations (1):
- An Nan Hospital, China Medical University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng CH, Cheng YY, Yuan MK, Juang YJ, Zeng XY, Chen CY, Foo NP. Impact of Personal Protective Equipment on Cardiopulmonary Resuscitation and Rescuer Safety. Emerg Med Int. 2023 Nov 30;2023:9697442. doi: 10.1155/2023/9697442. eCollection 2023. PMID 38077106